CLINICAL TRIAL: NCT06368596
Title: ENDS (ENDometriosis & FuSobacterium) Unveiling the Contribution of Fusobacterium Infection to the Development of Endometriosis
Acronym: ENDS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-04
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study arm (Other): Patients in reproductive age, who will undergo elective surgery for endometriosis.
  Interventions: Diagnostic Test: Fusobacterium detection
- Control arm (Other): Women in reproductive age, without endometriosis, as control group for secondary objective 1 and 2.
  Interventions: Diagnostic Test: Fusobacterium detection

INTERVENTIONS:
Diagnostic Test: Fusobacterium detection — One vaginal and one cervical swab will be collected from participants (both cases and controls) before surgery.
  During surgical intervention, routine biopsies of the endometriotic tissue will be done for all endometriosis types; further, small biopsies of apparently healthy endometrial tissue and of healthy peritoneum will be done, as per routine procedure.
  In the control group routine biopsies needed for the specific condition and small biopsies of endometrial tissue will be carried out.
  During these routine biopsies, a small additional quantity of tissue will be taken, which will be analyzed for the search for Fusobacterium.

SUMMARY:
This will be a clinical interventional longitudinal study, without pharmacological intervention/device evaluation.

A control group would however be recruited for secondary objective 1 and 2.

The study is classified as interventional, as Fusobacterium detection is not part of the routine management of these patients; from the patients' point of view, participation in the study will involve the execution of additional vaginal and cervical swabs as additional procedure, while the endometrial biopsy will not represent an additional examination, as the study will include only patients for whom this examination is expected as per normal clinical practice.

ELIGIBILITY:
Inclusion Criteria for study group:

* Age ≥ 18 years;
* endometriosis with clinical indication for either hysteroscopy or hysterectomy;
* signed informed consent to study participation and to personal data's treatment.

Inclusion Criteria for control group:

* need of elective gynecological surgery for causes other than endometriosis and malignancies;
* indication for hysteroscopy with endometrial biopsy;
* signed informed consent to study participation and to personal data's treatment.

Exclusion Criteria for both groups:

* lack of signed informed consent;
* Menopause
* antibiotic therapy in the 30 days before samples collection (including vaginal and cervical swab).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 845 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Fusobacterium sp presence (Y/N) in endometrial biopsy in women with endometriosis | At surgical intervention

SECONDARY OUTCOMES:
Fusobacterium presence (Y/N) in endometrial biopsy in women without endometriosis | At surgical intervention
Fusobacterium presence (Y/N) in vaginal and cervical swab in all women enrolled | At preoperative visit
Fusobacterium presence (Y/N) in endometrial biopsy in women with and without PID complicating endometriosis . | At surgical intervention
Fusobacterium presence (Y/N) in biopsies of endometrial tissue involving different sites (superficial lesions, deep endometriosis, ovarian endometrioma), if present | At surgical intervention
Fusobacterium presence (Y/N) in endometrial biopsy in women with and without infertility associated to endometriosis | At surgical intervention
Fusobacterium presence (Y/N) in endometrial biopsy in women with and without hysteroscopic signs of chronic endometritis in patients with and without endometriosis | At surgical intervention

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria di Negrar, Negrar, Verona, Italy